CLINICAL TRIAL: NCT04197050
Title: Effect of Sacubitril/Valsartan on Right Ventricular Dysfunctioning Patients With Connective Tissue Disease
Brief Title: Effect of Sacubitril/Valsartan on Reduced Right Ventricular Ejection Fraction in Patients With CTD
Acronym: EARLY-MYO-CTD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019-11-01R
Record Dates: First submitted 2019-11-27; First posted 2019-12-12 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2019-11

CONDITIONS: Myocardial Injury; Connective Tissue Diseases
Keywords: Connective Tissue Diseases; sacubitril/valsartan; Cardiovascular Magnetic Resonance; Extracellular Volume; exercise tolerance
MeSH Terms: conditions — Connective Tissue Diseases | interventions — sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sacubitril/valsartan group (Experimental): The diagnosis of CTD was made based on the clinical classification criteria. The patient was diagnosed by an echocardiography demonstration, when RVEF is suggested lower or equal to 45%, the patient will be considered a candidate after consent is signed. sacubitril/valsartan will be given.
  Interventions: Drug: Sacubitril / Valsartan Oral Tablet
- control group (No Intervention): The diagnosis of CTD was made based on the clinical classification criteria. The patient was diagnosed by an echocardiography demonstration, when RVEF is suggested lower or equal to 45%, the patient will be considered a candidate after consent is signed. Valsartan will be given.

INTERVENTIONS:
Drug: Sacubitril / Valsartan Oral Tablet — After recruiting participants and collecting the baseline information, sacubitril/valsartan group will receive sacubitril/valsartan and optimal pharmaceutical treatment (OPT). The control group will receive valsartan and OPT. A CMR scan and a post-processed imaging procedure will later be carried on in order to detect the cardiac impairment.
  Other Names: CMR examination
  Arms: sacubitril/valsartan group

SUMMARY:
Heart failure, one of the leading causes of connective tissue disease (CTD) mortality, has attracted increasing attention. Currently, no known study had focused on the effect of sacubitril/valsartan on right ventricular dysfunction and in the systemic disease induced heart disease. We aimed to observe the effect of sacubitril/valsartan on primary endpoints (6 minutes walking test and myocardial fibrosis) in CTD patients with right ventricular ejection fraction reduction (RV-HFrEF).

DETAILED DESCRIPTION:
Patients with CTD frequently exhibit multi-organ pathophysiological and functional damage. Heart failure, one of the leading causes of CTD mortality, has attracted increasing attention. Mostly, patients with CTD present with nonspecific cardiac symptoms, normal ECG, and preserved left ventricular ejection fraction (LVEF) and therefore do not receive an early cardiac diagnosis and treatment. Pulmonary arterial hypertension (PAH), right ventricular (RV) dilatation and hypertrophy might become the first and the most frequent cardiac findings. Sacubitril/valsartan, an angiotensin receptor-neprilysin inhibitors, is a "superstar" which inhibits both neprilysin and renin-angiotensin aldosterone system that closely related to the heart failure mechanism. It has been strongly recommended as class I drug in treating the patient with chronic HFrEF from 2017 ACC/AHA/HFSA heart failure guideline for the ability of dramatically reduce the cardiovascular mortality rate.

Cardiovascular magnetic resonance (CMR) is able to depict myocardial characteristics from structure to tissue properties using cine and late gadolinium enhancement (LGE) sequences. Newly developed imaging studies to date include T1 mapping and T1-derived extracellular volume estimation. All the previous studies in CTD have been restricted to patients with advanced cardiac involvement.

Together with clinical assessment and multi-imaging tests, the aim of the present study is going to observe the effect of sacubitril/valsartan on primary endpoints (6 minutes walking test and myocardial fibrosis) in CTD patients with RV-HFrEF.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-75 years old.
* confirmed CTD（including systemic lupus erythematosus, myositis, polymyositis, systemic sclerosis, sarcoid, Sjögren's syndrome or mixed connective tissue disease）
* SLEDAI ≤ 6 in patients with SLE or ESR ≤ 30 in patients with SSc
* already have OPT for CTD at least 3 month
* RVEF ≤ 45%
* Providing written informed consent

Exclusion Criteria:

* Documented coronary artery disease or prior angiography for coronary artery disease (>50% stenosis).
* Patients with known congenital heart disease or other systemic diseases that might induce RVrEF.
* Patients with standard metallic contraindications to CMR or an estimated glomerular filtration rate < 30 ml/min/1.73 m2.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-02-20 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Exercise tolerance | change between 1 and 6 months after treatment
  6 minutes walking test
Fibrosis Assessment | change between 1 and 6 months after treatment
  LGE assessment
Fibrosis Assessment | change between 1 and 6 months after treatment
  ECV quantification

SECONDARY OUTCOMES:
CTD activity | change between 1 and 6 months after treatment
  antinuclear antibody
Cardiovascular Mortality Rate | change between 1 and 6 months after treatment
  all cause of death

CONTACTS AND LOCATIONS:
Overall Officials: Meng Jiang, MD, Study Chair — RenJi Hospital, School of Medicine, Shanghai Jiantong University
Locations (1):
- Renji Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Braun J, Kruger K, Manger B, Schneider M, Specker C, Trappe HJ. Cardiovascular Comorbidity in Inflammatory Rheumatological Conditions. Dtsch Arztebl Int. 2017 Mar 24;114(12):197-203. doi: 10.3238/arztebl.2017.0197. PMID 28407841
- [Background] Leal GN, Silva KF, Franca CM, Lianza AC, Andrade JL, Campos LM, Bonfa E, Silva CA. Subclinical right ventricle systolic dysfunction in childhood-onset systemic lupus erythematosus: insights from two-dimensional speckle-tracking echocardiography. Lupus. 2015 May;24(6):613-20. doi: 10.1177/0961203314563135. Epub 2014 Dec 8. PMID 25492941
- [Background] Hassoun PM. The right ventricle in scleroderma (2013 Grover Conference Series). Pulm Circ. 2015 Mar;5(1):3-14. doi: 10.1086/679607. PMID 25992267
- [Background] Wigley FM, Lima JA, Mayes M, McLain D, Chapin JL, Ward-Able C. The prevalence of undiagnosed pulmonary arterial hypertension in subjects with connective tissue disease at the secondary health care level of community-based rheumatologists (the UNCOVER study). Arthritis Rheum. 2005 Jul;52(7):2125-32. doi: 10.1002/art.21131. PMID 15986394
- [Background] Argula RG, Karwa A, Lauer A, Gregg D, Silver RM, Feghali-Bostwick C, Schanpp LM, Egbert K, Usher BW, Ramakrishnan V, Hassoun PM, Strange C. Differences in Right Ventricular Functional Changes during Treatment between Systemic Sclerosis-associated Pulmonary Arterial Hypertension and Idiopathic Pulmonary Arterial Hypertension. Ann Am Thorac Soc. 2017 May;14(5):682-689. doi: 10.1513/AnnalsATS.201608-655OC. PMID 28282243
- [Background] Rich S, Pogoriler J, Husain AN, Toth PT, Gomberg-Maitland M, Archer SL. Long-term effects of epoprostenol on the pulmonary vasculature in idiopathic pulmonary arterial hypertension. Chest. 2010 Nov;138(5):1234-9. doi: 10.1378/chest.09-2815. PMID 21051399
- [Background] van de Veerdonk MC, Kind T, Marcus JT, Mauritz GJ, Heymans MW, Bogaard HJ, Boonstra A, Marques KM, Westerhof N, Vonk-Noordegraaf A. Progressive right ventricular dysfunction in patients with pulmonary arterial hypertension responding to therapy. J Am Coll Cardiol. 2011 Dec 6;58(24):2511-9. doi: 10.1016/j.jacc.2011.06.068. PMID 22133851
- [Background] Guo Q, Wu LM, Wang Z, Shen JY, Su X, Wang CQ, Gong XR, Yan QR, He Q, Zhang W, Xu JR, Jiang M, Pu J. Early Detection of Silent Myocardial Impairment in Drug-Naive Patients With New-Onset Systemic Lupus Erythematosus: A Three-Center Prospective Study. Arthritis Rheumatol. 2018 Dec;70(12):2014-2024. doi: 10.1002/art.40671. PMID 30070061
- [Background] Owens AT, Brozena S, Jessup M. Neprilysin Inhibitors: Emerging Therapy for Heart Failure. Annu Rev Med. 2017 Jan 14;68:41-49. doi: 10.1146/annurev-med-052915-015509. Epub 2016 Sep 21. PMID 27686019
- [Background] McMurray JJ, Packer M, Desai AS, Gong J, Lefkowitz MP, Rizkala AR, Rouleau JL, Shi VC, Solomon SD, Swedberg K, Zile MR; PARADIGM-HF Investigators and Committees. Angiotensin-neprilysin inhibition versus enalapril in heart failure. N Engl J Med. 2014 Sep 11;371(11):993-1004. doi: 10.1056/NEJMoa1409077. Epub 2014 Aug 30. PMID 25176015
- [Background] Yancy CW, Jessup M, Bozkurt B, Butler J, Casey DE Jr, Colvin MM, Drazner MH, Filippatos GS, Fonarow GC, Givertz MM, Hollenberg SM, Lindenfeld J, Masoudi FA, McBride PE, Peterson PN, Stevenson LW, Westlake C. 2017 ACC/AHA/HFSA Focused Update of the 2013 ACCF/AHA Guideline for the Management of Heart Failure: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines and the Heart Failure Society of America. Circulation. 2017 Aug 8;136(6):e137-e161. doi: 10.1161/CIR.0000000000000509. Epub 2017 Apr 28. No abstract available. PMID 28455343
- [Background] Ponikowski P, Voors AA, Anker SD, Bueno H, Cleland JGF, Coats AJS, Falk V, Gonzalez-Juanatey JR, Harjola VP, Jankowska EA, Jessup M, Linde C, Nihoyannopoulos P, Parissis JT, Pieske B, Riley JP, Rosano GMC, Ruilope LM, Ruschitzka F, Rutten FH, van der Meer P; ESC Scientific Document Group. 2016 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: The Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC)Developed with the special contribution of the Heart Failure Association (HFA) of the ESC. Eur Heart J. 2016 Jul 14;37(27):2129-2200. doi: 10.1093/eurheartj/ehw128. Epub 2016 May 20. No abstract available. PMID 27206819
- [Background] Velazquez EJ, Morrow DA, DeVore AD, Duffy CI, Ambrosy AP, McCague K, Rocha R, Braunwald E; PIONEER-HF Investigators. Angiotensin-Neprilysin Inhibition in Acute Decompensated Heart Failure. N Engl J Med. 2019 Feb 7;380(6):539-548. doi: 10.1056/NEJMoa1812851. Epub 2018 Nov 11. PMID 30415601
- [Background] Pascual-Figal D, Wachter R, Senni M, Belohlavek J, Noe A, Carr D, Butylin D. Rationale and design of TRANSITION: a randomized trial of pre-discharge vs. post-discharge initiation of sacubitril/valsartan. ESC Heart Fail. 2018 Apr;5(2):327-336. doi: 10.1002/ehf2.12246. Epub 2017 Dec 14. PMID 29239515
- [Background] Jiang M, Wang Z, Su X, Gong X, Pu J, Wu L, Liu C, Yao Q, Kong L, Xu J, He B. The Significance of Interstitial Fibrosis on Left Ventricular Function in Hypertensive versus Hypertrophic Cardiomyopathy. Sci Rep. 2018 Jul 3;8(1):9995. doi: 10.1038/s41598-018-27049-1. PMID 29968754
- [Background] Jiang M, Xu J, He B. Diffuse Epicardial Involvement on Cardiac Magnetic Resonance Imaging. JAMA Cardiol. 2016 Oct 1;1(7):845-846. doi: 10.1001/jamacardio.2016.2557. No abstract available. PMID 27579709
- [Background] Jiang M, Pu J, Yao J, Xu J, He B. An acromegaly-induced cardiomyopathy mimicking amyloidosis: (Manifestation of acromegaly-induced-cardiomyopathy). Int J Cardiol. 2016 Jul 15;215:60-1. doi: 10.1016/j.ijcard.2016.04.043. Epub 2016 Apr 13. No abstract available. PMID 27111161
- [Background] Leng S, Jiang M, Zhao XD, Allen JC, Kassab GS, Ouyang RZ, Tan JL, He B, Tan RS, Zhong L. Three-Dimensional Tricuspid Annular Motion Analysis from Cardiac Magnetic Resonance Feature-Tracking. Ann Biomed Eng. 2016 Dec;44(12):3522-3538. doi: 10.1007/s10439-016-1695-2. Epub 2016 Jul 19. PMID 27436293
- [Background] Wu LM, An DL, Yao QY, Ou YZ, Lu Q, Jiang M, Xu JR. Hypertrophic cardiomyopathy and left ventricular hypertrophy in hypertensive heart disease with mildly reduced or preserved ejection fraction: insight from altered mechanics and native T1 mapping. Clin Radiol. 2017 Oct;72(10):835-843. doi: 10.1016/j.crad.2017.04.019. Epub 2017 May 25. PMID 28552325